CLINICAL TRIAL: NCT04191798
Title: Randomized Study of the KinexConnect Telerehabilitation System Versus Outpatient Physical Therapy After Total Knee Arthroplasty
Brief Title: Study of the KinexConnect Telerehabilitation System (KCTRS)
Acronym: KCTRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kinex Medical Company, LLC (Industry)
Collaborators: Health Factors Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KC-07
Record Dates: First submitted 2019-12-04; First posted 2019-12-10 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Osteoarthritis, Knee
Keywords: Arthroplasty; Knee Replacement; Rehab at home; Virtual PT; Remote Patient Monitoring; Patient Engagement; TKR; TKA
MeSH Terms: conditions — Osteoarthritis, Knee; Patient Participation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All TUG and RoM assessments will be performed by trained physician assistants who will remain blinded to allocation throughout the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KinexConnect (Experimental): Rehab at Home Patients
  Interventions: Behavioral: Telerehabilitation using the KinexConnect system for rehabilitation after TKA.
- Outpatient PT (Active Comparator): In-person PT patients
  Interventions: Behavioral: Traditional outpatient PT for rehabilitation after TKA.

INTERVENTIONS:
Behavioral: Telerehabilitation using the KinexConnect system for rehabilitation after TKA. — KinexConnect subjects are asked to Perform CPM therapy for 4 weeks. Perform a KCK home exercise program (HEP) for 6 weeks.
  Arms: KinexConnect
Behavioral: Traditional outpatient PT for rehabilitation after TKA. — Control subjects are asked to undergo standard outpatient physical therapy (PT) with a licensed physical therapist plus supplemental home exercises as directed. Nominally patients are expected to have 3 PT sessions per week for 4 weeks.
  Arms: Outpatient PT

SUMMARY:
A randomized, single-blind study comparing telerehabilitation at home with continuous passive motion (CPM) and a tablet-based patient engagement application (KinexConnect) versus traditional outpatient physical therapy (PT) following total knee arthroplasty (TKA).

DETAILED DESCRIPTION:
The Randomized Study of the KinexConnect Telerehabilitation System is a 1:1 randomized, single-blind, prospective cohort study to be conducted at one investigational site in the United States. The study compares at-home telerehabilitation system versus traditional outpatient PT following total knee arthroplasty (TKA). The telerehabilitation system involves a tablet-enabled patient engagement application, the KinexConnect App, to be used in conjunction with a continuous passive motion (CPM) machine.

ELIGIBILITY:
Inclusion Criteria:

1. Planned for a primary unilateral TKA.
2. At least 21 years of age.
3. Capable of understanding the study requirements and giving written informed consent.
4. Willing and able to comply with either therapy program.
5. Has easy access to caregiver support.

Exclusion Criteria:

1. Active range-of-motion (ARoM) < 80 degrees in target knee.
2. Unable to read and write in English.
3. Lack of email capability to receive recovery trend information.
4. Previous knee intervention in target knee.
5. Previous knee joint infection in either knee.
6. Received a revision TKA (opposite knee).
7. Planned for bilateral TKA.
8. Self-reported pregnancy.
9. Reason for arthroplasty being for the treatment of fracture, infection or malignancy.
10. Other physical or mental impairments or medical conditions that may affect ability to complete therapy as prescribed.
11. Unwilling to participate.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Timed up and Go (TUG) Test score | 3 months
  The TUG score is the measurement of time for a person to rise from a standard armchair (seat height 46 cm), walk 3 meters, turn, walk back to the chair, and sit down as quickly as possible. The mean scores for patients in both arms are derived and compared against each other. Closer the trial arm mean is to the control arm mean, the better.
Change in the Timed up and Go (TUG) Test score | 1 year
  The TUG score is the measurement of time for a person to rise from a standard armchair (seat height 46 cm), walk 3 meters, turn, walk back to the chair, and sit down as quickly as possible. The mean scores for patients in both arms are derived and compared against each other. Closer the trial arm mean is to the control arm mean, the better.
Economic Benefit | 3 months
  Expenses associated with rehabilitation after surgery will be based on costs associated with CPM rental fees and outpatient physical therapy visits. Estimates will be applied wherever actual expense data is not available.
Economic Benefit | 1 year
  Expenses associated with rehabilitation after surgery will be based on costs associated with CPM rental fees and outpatient physical therapy visits. Estimates will be applied wherever actual expense data is not available.

SECONDARY OUTCOMES:
Change in Active Range of Motion (ARoM) | 3 months and 6 months
  Active Range of Motion is the difference between the maximum Flexion and maximum Extension the patient is able to achieve with independent effort
Change in Passive Range of Motion (PRoM) | 3 months and 6 months
  Passive Range of Motion is the difference between the maximum Flexion and maximum Extension the patient is able to achieve when bearable force is exerted by the clinician.
Change in Pain as measured by the Verbal Descriptive Scale (VDS) | 3 months and 1 year
  This is a self reported outcome by the patient based on their expression of pain at a given time point when presented with the 7 verbal cues.
  The levels of pain reported vary from "No Pain" to "Most Intense Pain Imaginable". Higher the intensity of pain, worse the outcome
Change in the Knee Osteoarthritis Outcome Score (KOOS) | 3 months and 1 year
  The KOOS is a standardized and validated patient outcome score that assess functional limitation in patient with knee osteoarthritis. The survey questionnaire is filled out in its entirety by the patient.
  The five patient-relevant subscales of KOOS are scored separately: Pain (nine items); Symptoms (seven items); ADL Function (17 items); Sport and Recreation Function (five items); Quality of Life (four items). A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Change in the New Knee Society Score (NKSS) - Patient Satisfaction and Expectation | 3 months and 1 year
  The patient satisfaction and patient expectation scores are calculated by having the relevant sections of the survey questionnaire is filled out in its entirety by the patient.
  Patient Satisfaction is scored 0 - 40 points and Patient Expectation is scored 0 -15 points. with Zero being the worst outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Barron Bremner, DO, Principal Investigator — Des Moines Orthopedic Suregons
Locations (1):
- Des Moines Orthopedic Surgeons, Des Moines, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pastora-Bernal JM, Martin-Valero R, Baron-Lopez FJ, Estebanez-Perez MJ. Evidence of Benefit of Telerehabitation After Orthopedic Surgery: A Systematic Review. J Med Internet Res. 2017 Apr 28;19(4):e142. doi: 10.2196/jmir.6836. PMID 28455277
- [Background] Shukla H, Nair SR, Thakker D. Role of telerehabilitation in patients following total knee arthroplasty: Evidence from a systematic literature review and meta-analysis. J Telemed Telecare. 2017 Feb;23(2):339-346. doi: 10.1177/1357633X16628996. Epub 2016 Jul 9. PMID 26843466
- [Background] Jiang S, Xiang J, Gao X, Guo K, Liu B. The comparison of telerehabilitation and face-to-face rehabilitation after total knee arthroplasty: A systematic review and meta-analysis. J Telemed Telecare. 2018 May;24(4):257-262. doi: 10.1177/1357633X16686748. Epub 2016 Dec 27. PMID 28027679
- [Background] Kline PW, Melanson EL, Sullivan WJ, Blatchford PJ, Miller MJ, Stevens-Lapsley JE, Christiansen CL. Improving Physical Activity Through Adjunct Telerehabilitation Following Total Knee Arthroplasty: Randomized Controlled Trial Protocol. Phys Ther. 2019 Jan 1;99(1):37-45. doi: 10.1093/ptj/pzy119. PMID 30329126
- [Background] Ong KL, Lotke PA, Lau E, Manley MT, Kurtz SM. Prevalence and Costs of Rehabilitation and Physical Therapy After Primary TJA. J Arthroplasty. 2015 Jul;30(7):1121-6. doi: 10.1016/j.arth.2015.02.030. Epub 2015 Feb 28. PMID 25765130
- [Result] Rondon AJ, Phillips JLH, Fillingham YA, Gorica Z, Austin MS, Courtney PM. Bundled Payments Are Effective in Reducing Costs Following Bilateral Total Joint Arthroplasty. J Arthroplasty. 2019 Jul;34(7):1317-1321.e2. doi: 10.1016/j.arth.2019.03.041. Epub 2019 Mar 28. PMID 30992236
- [Result] Bini SA, Mahajan J. Clinical outcomes of remote asynchronous telerehabilitation are equivalent to traditional therapy following total knee arthroplasty: A randomized control study. J Telemed Telecare. 2017 Feb;23(2):239-247. doi: 10.1177/1357633X16634518. Epub 2016 Jul 9. PMID 26940798
- [Result] Moffet H, Tousignant M, Nadeau S, Merette C, Boissy P, Corriveau H, Marquis F, Cabana F, Ranger P, Belzile EL, Dimentberg R. In-Home Telerehabilitation Compared with Face-to-Face Rehabilitation After Total Knee Arthroplasty: A Noninferiority Randomized Controlled Trial. J Bone Joint Surg Am. 2015 Jul 15;97(14):1129-41. doi: 10.2106/JBJS.N.01066. PMID 26178888
- [Result] Correia FD, Nogueira A, Magalhaes I, Guimaraes J, Moreira M, Barradas I, Teixeira L, Tulha J, Seabra R, Lains J, Bento V. Home-based Rehabilitation With A Novel Digital Biofeedback System versus Conventional In-person Rehabilitation after Total Knee Replacement: a feasibility study. Sci Rep. 2018 Jul 26;8(1):11299. doi: 10.1038/s41598-018-29668-0. PMID 30050087
- [Result] Correia FD, Nogueira A, Magalhaes I, Guimaraes J, Moreira M, Barradas I, Molinos M, Teixeira L, Tulha J, Seabra R, Lains J, Bento V. Medium-Term Outcomes of Digital Versus Conventional Home-Based Rehabilitation After Total Knee Arthroplasty: Prospective, Parallel-Group Feasibility Study. JMIR Rehabil Assist Technol. 2019 Feb 28;6(1):e13111. doi: 10.2196/13111. PMID 30816849
- [Result] Fleischman AN, Crizer MP, Tarabichi M, Smith S, Rothman RH, Lonner JH, Chen AF. 2018 John N. Insall Award: Recovery of Knee Flexion With Unsupervised Home Exercise Is Not Inferior to Outpatient Physical Therapy After TKA: A Randomized Trial. Clin Orthop Relat Res. 2019 Jan;477(1):60-69. doi: 10.1097/CORR.0000000000000561. PMID 30794229
- [Result] Moffet H, Tousignant M, Nadeau S, Merette C, Boissy P, Corriveau H, Marquis F, Cabana F, Belzile EL, Ranger P, Dimentberg R. Patient Satisfaction with In-Home Telerehabilitation After Total Knee Arthroplasty: Results from a Randomized Controlled Trial. Telemed J E Health. 2017 Feb;23(2):80-87. doi: 10.1089/tmj.2016.0060. Epub 2016 Aug 16. PMID 27529575
- [Result] Tousignant M, Moffet H, Nadeau S, Merette C, Boissy P, Corriveau H, Marquis F, Cabana F, Ranger P, Belzile EL, Dimentberg R. Cost analysis of in-home telerehabilitation for post-knee arthroplasty. J Med Internet Res. 2015 Mar 31;17(3):e83. doi: 10.2196/jmir.3844. PMID 25840501
- [Result] Buhagiar MA, Naylor JM, Harris IA, Xuan W, Kohler F, Wright R, Fortunato R. Effect of Inpatient Rehabilitation vs a Monitored Home-Based Program on Mobility in Patients With Total Knee Arthroplasty: The HIHO Randomized Clinical Trial. JAMA. 2017 Mar 14;317(10):1037-1046. doi: 10.1001/jama.2017.1224. PMID 28291891
- See also: SURGICAL MANAGEMENT OF OSTEOARTHRITIS OF THE KNEE EVIDENCE-BASED CLINICAL PRACTICE GUIDELINE — http://www.orthoguidelines.org/topic?id=1019